CLINICAL TRIAL: NCT04847726
Title: Perfluorobutane-enhanced Ultrasound as a Diagnostic Tool for Hepatocellular Carcinoma in Individuals With High Risk: Intraindividual Comparison With Sulfur Hexafluoride-enhanced Ultrasound
Brief Title: Contrast-enhanced Ultrasound With Perfluorobutane and Sulfur Hexafluoride for Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUH-1807-166
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; Contrast-enhanced ultrasound; Perfluorobutane; Sulfur hexafluoride
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Study participants underwent contrast-enhanced ultrasound with perfluorobutane and sulfur hexafluoride. The diagnostic performance will be compared intra-individually.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CEUS with perfluorobutane and sulfur hexafluoride (Experimental): Contrast-enhanced ultrasound with perfluorobutane and sulfur hexafluoride for the hepatic lesion.
  Interventions: Diagnostic Test: contrast enhanced ultrasound; Diagnostic Test: Dynamic CT; Diagnostic Test: Liver MRI

INTERVENTIONS:
Diagnostic Test: contrast enhanced ultrasound — contrast enhanced ultrasound with perfluorobutane and sulfur hexafluoride
Diagnostic Test: Dynamic CT — Participants underwent dynamic CT for hepatic lesion
Diagnostic Test: Liver MRI — Participants underwent liver MRI for hepatic lesion

SUMMARY:
Intra-individual comparison of diagnostic performance of CEUS With perfluorobutane and sulfur hexafluoride for HCC in high-risk Individuals, and their role in the diagnostic algorithm of HCC.

DETAILED DESCRIPTION:
The investigators would compare the diagnostic performance for HCC at high-risk individuals between both USG contrast agents.

ELIGIBILITY:
Inclusion Criteria:

* high-risk for HCC (liver cirrhosis, chronic hepatitis B)
* treatment-naive hepatic nodule (>= 1cm) on preceding CT, MR or ultrasound

Exclusion Criteria:

* severe cardiopulmonary dysfunction
* pregnancy
* refusal to enroll study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy for HCC: non-inferiority test | up to 3 months
  The per-lesion diagnostic accuracy for HCC of CEUS with perfluorobutane and sulfur hexafluoride using the same diagnostic criteria (arterial phase hyperenehancement with mild and late (≥ 60 sec) washout).

SECONDARY OUTCOMES:
Diagnostic performance of perfulorobutane enhanced USG using different definition of washout | up to 3 months
  Per-lesion sensitivity and specificity for diagnosing HCC using different time windows for assessing washout in PFB-US

OTHER OUTCOMES:
Role of perfluorobutane enhanced USG in EASL diagnostic algorithm of HCC | up to 3 months
  The number of perfluorobutane enhanced USG diagnosed HCC that were missed by prior gadoxetic-acid MRI to simulate diagnostic algorithm for HCC and reveal the role of PFB-US as a second-line diagnostic modality

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, Dr., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

REFERENCES:
- [Derived] Kang HJ, Lee JM, Yoon JH, Yoo J, Choi Y, Joo I, Han JK. Sonazoid versus SonoVue(R) for Diagnosing Hepatocellular Carcinoma Using Contrast-Enhanced Ultrasound in At-Risk Individuals: A Prospective, Single-Center, Intraindividual, Noninferiority Study. Korean J Radiol. 2022 Nov;23(11):1067-1077. doi: 10.3348/kjr.2022.0388. Epub 2022 Sep 30. PMID 36196767